CLINICAL TRIAL: NCT02477592
Title: A Prospective Randomized Study of a Novel Individualized Substrate Modification Approach Versus Stepwise Ablation for the Treatment of Long-standing Persistent Atrial Fibrillation
Brief Title: a Novel Individualized Substrate Modification Approach for the Treatment of Long-standing Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 仁济伦审[2014]116K
Record Dates: First submitted 2015-06-08; First posted 2015-06-23 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-01

CONDITIONS: Atrial Fibrillation
Keywords: long standing persistent atrial fibrillation; novel approach; ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individualized substrate modification (Experimental): Circumferential pulmonary vein isolation(CPVI) ablation and left atrial roof linear ablation first,then substrate mapping in sinus rhythm followed by Individualized substrate modification.
  Interventions: Procedure: individualized substrate modification
- Stepwise ablation (Active Comparator): CPVI ablation,left atrial roof linear ablation,mitral isthmus linear ablation,complex fractionated atrial electrograms ablation step by step.
  Interventions: Procedure: stepwise ablation

INTERVENTIONS:
Procedure: individualized substrate modification — CPVI ablation and left atrial roof linear ablation first,then substrate mapping in sinus rhythm followed by individualized substrate modification.
  Arms: Individualized substrate modification
Procedure: stepwise ablation — CPVI ablation,left atrial roof linear ablation,mitral isthmus linear ablation,complex fractionated atrial electrograms ablation step by step.
  Arms: Stepwise ablation

SUMMARY:
The purpose of this study is to compare effectiveness of two substrate modification approaches in long-standing persistent atrial fibrillation patients, and hypothesized that a substrate-based, individualized substrate modification (ISM)approach should be superior to traditional stepwise ablation(SA). To the best of investigator's knowledge, this was the first study to evaluate the "real" substrate by means of electro-anatomic mapping and to perform "true" substrate modification in long standing persistent atrial fibrillation ablation(LPAF).

DETAILED DESCRIPTION:
Catheter ablation (CA) is highly effective for paroxysmal atrial fibrillation(AF), it is modestly effective for long standing persistent atrial fibrillation ablation(LPAF) even with complex or combined approaches, which is mainly attributed to the substrate underlying AF remodeling. Severity of atrial fibrosis is closely associated with clinical outcomes after CA for AF . The more atrial scars and fibrosis present, the lower the success rate for AF ablation. Patients with LPAF have many more areas with scars and fibrosis than those with paroxysmal AF or non-AF controls. The MRI delayed enhancement technique provides a non-interventional tool for evaluation of atrial fibrosis, however, it must be performed in sinus rhythm.Three-dimensional electro anatomic mapping has proven as accurate as MRI and can be performed easily during AF ablation, thus providing a good tool for evaluation of atrial substrate during LPAF ablation.

Although electro-anatomic mapping provided a desirable surrogate for delayed enhancement MRI to define AF substrate, there was an important technical issue to be considered. There were no good techniques to predict a desirable tip-tissue contact before the contact force catheter was applied. A poor tip-tissue contact could render the results of voltage mapping less reliable. On the other hand, excessively high contact force could increase the risk of steam pop and cardiac perforation during ablation. Hence it was important to use the contact force catheter to perform substrate mapping and ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 72years
* History of LPAF for ≥1 and ≤ 5 years
* Written informed consent provided
* Acceptance of catheter ablation treatment
* Acceptance of post-ablation follow-up

Exclusion Criteria:

* Prior history of catheter ablation or surgical ablation
* Abnormal coagulation; contraindication for anti-coagulation
* left atrium diameter ≥ 55mm
* left atrium thrombus

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
atrial fibrillation free rate on or off antiarrhythmic drugs (AADs) after initial ablation | 1 year

SECONDARY OUTCOMES:
Number of participants with adverse event | 1 year
  pericardial tamponade and thromboembolism event
Prevalence of recurrent atrial flutter | 1 year
Proportion of pulmonary vein isolation | 1 year
Proportion of acute pulmonary vein re-connection | 1 year
Fluoroscopy exposure time | 1 year
Total ablation time | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xinhua Wang, MD,PHD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiaotong University school of medicine,Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.e21. doi: 10.1016/j.hrthm.2011.12.016. Epub 2012 Mar 1. No abstract available. PMID 22386883
- [Result] Camm AJ, Lip GY, De Caterina R, Savelieva I, Atar D, Hohnloser SH, Hindricks G, Kirchhof P; ESC Committee for Practice Guidelines (CPG). 2012 focused update of the ESC Guidelines for the management of atrial fibrillation: an update of the 2010 ESC Guidelines for the management of atrial fibrillation. Developed with the special contribution of the European Heart Rhythm Association. Eur Heart J. 2012 Nov;33(21):2719-47. doi: 10.1093/eurheartj/ehs253. Epub 2012 Aug 24. No abstract available. PMID 22922413
- [Result] Chao TF, Tsao HM, Lin YJ, Tsai CF, Lin WS, Chang SL, Lo LW, Hu YF, Tuan TC, Suenari K, Li CH, Hartono B, Chang HY, Ambrose K, Wu TJ, Chen SA. Clinical outcome of catheter ablation in patients with nonparoxysmal atrial fibrillation: results of 3-year follow-up. Circ Arrhythm Electrophysiol. 2012 Jun 1;5(3):514-20. doi: 10.1161/CIRCEP.111.968032. Epub 2012 May 1. PMID 22550126
- [Result] Brooks AG, Stiles MK, Laborderie J, Lau DH, Kuklik P, Shipp NJ, Hsu LF, Sanders P. Outcomes of long-standing persistent atrial fibrillation ablation: a systematic review. Heart Rhythm. 2010 Jun;7(6):835-46. doi: 10.1016/j.hrthm.2010.01.017. Epub 2010 Jan 22. PMID 20206320
- [Result] Sawhney N, Anousheh R, Chen W, Feld GK. Circumferential pulmonary vein ablation with additional linear ablation results in an increased incidence of left atrial flutter compared with segmental pulmonary vein isolation as an initial approach to ablation of paroxysmal atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Jun;3(3):243-8. doi: 10.1161/CIRCEP.109.924878. Epub 2010 Mar 25. PMID 20339034
- [Result] Sawhney N, Anand K, Robertson CE, Wurdeman T, Anousheh R, Feld GK. Recovery of mitral isthmus conduction leads to the development of macro-reentrant tachycardia after left atrial linear ablation for atrial fibrillation. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):832-7. doi: 10.1161/CIRCEP.111.964817. Epub 2011 Sep 30. PMID 21965530
- [Result] Chen M, Yang B, Chen H, Ju W, Zhang F, Tse HF, Cao K. Randomized comparison between pulmonary vein antral isolation versus complex fractionated electrogram ablation for paroxysmal atrial fibrillation. J Cardiovasc Electrophysiol. 2011 Sep;22(9):973-81. doi: 10.1111/j.1540-8167.2011.02051.x. Epub 2011 May 3. PMID 21539635
- [Result] Verma A, Wazni OM, Marrouche NF, Martin DO, Kilicaslan F, Minor S, Schweikert RA, Saliba W, Cummings J, Burkhardt JD, Bhargava M, Belden WA, Abdul-Karim A, Natale A. Pre-existent left atrial scarring in patients undergoing pulmonary vein antrum isolation: an independent predictor of procedural failure. J Am Coll Cardiol. 2005 Jan 18;45(2):285-92. doi: 10.1016/j.jacc.2004.10.035. PMID 15653029
- [Result] Mahnkopf C, Badger TJ, Burgon NS, Daccarett M, Haslam TS, Badger CT, McGann CJ, Akoum N, Kholmovski E, Macleod RS, Marrouche NF. Evaluation of the left atrial substrate in patients with lone atrial fibrillation using delayed-enhanced MRI: implications for disease progression and response to catheter ablation. Heart Rhythm. 2010 Oct;7(10):1475-81. doi: 10.1016/j.hrthm.2010.06.030. Epub 2010 Jul 1. PMID 20601148
- [Result] Teh AW, Kistler PM, Lee G, Medi C, Heck PM, Spence SJ, Sparks PB, Morton JB, Kalman JM. Electroanatomic remodeling of the left atrium in paroxysmal and persistent atrial fibrillation patients without structural heart disease. J Cardiovasc Electrophysiol. 2012 Mar;23(3):232-8. doi: 10.1111/j.1540-8167.2011.02178.x. Epub 2011 Sep 28. PMID 21955090
- [Result] Oakes RS, Badger TJ, Kholmovski EG, Akoum N, Burgon NS, Fish EN, Blauer JJ, Rao SN, DiBella EV, Segerson NM, Daccarett M, Windfelder J, McGann CJ, Parker D, MacLeod RS, Marrouche NF. Detection and quantification of left atrial structural remodeling with delayed-enhancement magnetic resonance imaging in patients with atrial fibrillation. Circulation. 2009 Apr 7;119(13):1758-67. doi: 10.1161/CIRCULATIONAHA.108.811877. Epub 2009 Mar 23. PMID 19307477
- [Result] Park JH, Pak HN, Choi EJ, Jang JK, Kim SK, Choi DH, Choi JI, Hwang C, Kim YH. The relationship between endocardial voltage and regional volume in electroanatomical remodeled left atria in patients with atrial fibrillation: comparison of three-dimensional computed tomographic images and voltage mapping. J Cardiovasc Electrophysiol. 2009 Dec;20(12):1349-56. doi: 10.1111/j.1540-8167.2009.01557.x. PMID 19602027